CLINICAL TRIAL: NCT00315614
Title: Islet Cell Transplantation Alone and CD34+ Enriched Donor Bone Marrow Cell Infusion in Patients With Type 1 Diabetes Mellitus; Steroid Free Regimen
Brief Title: Islet Cell Transplantation Alone and CD34+ Donor Bone Marrow Cell Infusion in Type 1 Diabetes Mellitus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: We did not achieve a tolerogenic profile. Subjects withdrew from protocol and enrolled in other islet transplant trials.
Sponsor: University of Miami (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Diabetes Research Institute Foundation (Other)
Responsible Party: Principal Investigator, Rodolfo Alejandro, Professor of Medicine, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000/0024; R01DK056953 (NIH)
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Results first posted 2014-02-10 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Islet Transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Islets of Langerhans Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Islet Transplantation and Bone Marrow (Experimental): Administration of islets and infusion of CD34 enriched Bone Marrow cells in subjects with type 1 diabetes, impaired awareness of hypoglycemia and severe hypoglycemia.
  Interventions: Biological: Islet Transplantation and Bone Marrow

INTERVENTIONS:
Biological: Islet Transplantation and Bone Marrow — Islet transplantation and CD34 Bone Marrow infusion in subjects with type 1 diabetes.
  Other Names: Islet; type 1 DM; Bone marrow

SUMMARY:
SPECIFIC AIMS:

* To reverse hyperglycemia and insulin dependency in patients with Type 1 diabetes mellitus by islet cell transplantation.
* To induce a state of donor specific tolerance and eliminate the need for continuous immunosuppressive therapy by simultaneous transplantation of donor bone marrow cells with islets and utilization of the monoclonal antibody Campath-1H for induction of Immunosuppression.
* To assess long-term function of successful islet cell transplants in patients with Type 1 diabetes mellitus.
* To determine whether the natural history of the microvascular, macrovascular and neuropathic complications are altered following successful transplantation of islet

DETAILED DESCRIPTION:
In our current protocol (IRB #2000/0024) the immunosuppressive regimen, comprised of induction with daclizumab and maintenance therapy with sirolimus and tacrolimus, has been combined with the infusion of CD34+ enriched donor bone marrow stem cells in an attempt to create a chimeric state and hence induce donor tolerance. This strategy was tested by evaluating graft survival following the removal of all immunosuppressive medication after one year.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18 and 65 years of age
2. Patients with type 1 diabetes mellitus for more than 5 years duration
3. One or more of the following:

   * Hypoglycemia unawareness - judged by history of blood sugars <54 on glucometer without symptoms and/or hypoglycemic episodes requiring assistance from either family, glucagon administration or emergency services
   * Poor diabetes control (HbA1c>8% or >2 visits/yr to hospital for treatment of ketoacidosis) despite intensive insulin therapy
   * Progressive complications of type 1 diabetes mellitus
4. Body Mass Index (BMI) ≤26

Exclusion Criteria:

1. Untreated proliferative diabetic retinopathy;
2. HbA1C > 12%;
3. Insulin requirement > 1.0u/kg/d
4. Stimulated or basal C-peptide > 0.3 ng/ml
5. Creatinine clearance < 60 and/or serum creatinine consistently > 1.5mg/dl;
6. Macroalbuminuria > 300mg albumin in 24 hours
7. Presence of panel reactive antibodies > 20%;
8. Previous/concurrent organ transplantation (except failed islet cell transplantation);
9. Any medical condition requiring chronic use of steroids;
10. Malignancy or previous malignancy (except non-melanomatous skin cancer);
11. X-ray evidence of pulmonary infection;
12. Active infections;
13. Positive tuberculin test (unless proof of adequate treatment for latent tuberculosis can be provided)
14. Active peptic ulcer disease,
15. Gall stones and/or portal hypertension and/or hemangioma on liver ultrasound;
16. Serological evidence of HIV, HBV (HBsAg+ and/or HBcAb+ and/or HBsAb+ without evidence of vaccination), HTLV-1 or HCV;
17. Negative serology for Epstein Barr virus (EBV) or evidence of acute infection (IgM>IgG);
18. Abnormal liver function test;
19. Anemia (hemoglobin <12.0 g/dl);
20. Hyperlipidemia (fasting total cholesterol >240mg/dl and/or fasting triglycerides >200mg/dl and/or fasting LDL cholesterol>140mg/dl);
21. Body Mass Index above 26 and/or weight >80kg;
22. Prostate specific antigen (PSA) > 4 ng/ml;
23. Unstable cardiovascular status (including positive stress echocardiography if >age 35);
24. Active alcohol or substance abuse;
25. Sexually active females who are not: a) post-menopausal, b) surgically sterile, or c) not using an acceptable method of contraception (oral contraceptives, Norplant, Depo-Provera, and barrier devices are acceptable; condoms used alone are not acceptable);
26. Positive pregnancy test or intent for future pregnancy, or male subject's intent to procreate.
27. Any condition or any circumstances that makes it unsafe to undergo an islet cell transplant.
28. History of previous transplant or previous bone marrow infusion.
29. Persistent leucopenia (white blood cell count <3,000/mm3

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2000-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Alejandro, MD, Principal Investigator — Diabetes Research Institute University of Miami
Locations (1):
- Diabetes Research Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Single arm few subjects.

REFERENCES:
- [Derived] Tharavanij T, Betancourt A, Messinger S, Cure P, Leitao CB, Baidal DA, Froud T, Ricordi C, Alejandro R. Improved long-term health-related quality of life after islet transplantation. Transplantation. 2008 Nov 15;86(9):1161-7. doi: 10.1097/TP.0b013e31818a7f45. PMID 19005394
- See also: Diabetes Research Institute web site — http://www.diabetesresearch.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Islet Transplantation and Bone Marrow: Islet transplantation and CD34 Bone Marrow infusion in subjects with type 1 diabetes, impaired hypoglycemia awareness and severe hypoglycemia.
Period: Overall Study
Arm/Group | Islet Transplantation and Bone Marrow
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Islet Transplantation and CD34 Bone Marrow: Islet Transplantation: Islet transplantation
Arm/Group | Islet Transplantation and CD34 Bone Marrow
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: The Achievement of Persistent Islet Function Following Cessation of Immunosuppression.
Description: Immunosuppression was never discontinued. Patients elected to move to other trials to receive additional islet infusions. Since immunosuppression was never discontinued we were not able to evaluate the primary endpoint.
Time Frame: for the duration of islet graft function
Population: IImmunosuppression was never discontinued. Patients elected to move to other trials to receive additional islet infusions. Since immunosuppression was never discontinued we were not able to evaluate the primary endpoint. No data available to analyze.
Arm/Group | Islet Transplantation and CD34 Bone Marrow
Number analyzed (Participants) | 0
Value | 0

2. Primary Outcome: A Reduction or Absence of Rejection Episodes
Description: Number of rejection episodes after transplantation. Immunosuppression was never discontinued. Patients elected to move to other trials to receive additional islet infusions. Since immunosuppression was never discontinued we were not able to evaluate the primary endpoint.
Time Frame: for the duration of islet graft function
Population: as for outcome 1
Arm/Group | Islet Transplantation and Bone Marrow
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Subjects With Basal C-peptide Greater Than 0.5 ng/ml
Description: Number of subjects with basal C-peptide greater than 0.5 ng/ml prior to weaning of immunosuppression;
Time Frame: for the duration of islet graft function
Measure: Count of Participants; unit: Participants
Arm/Group | Islet Transplantation and Bone Marrow
Number analyzed (Participants) | 3
Participants | 3

4. Secondary Outcome: Number of Subjects With Reduction of Severe Hypoglycemia and Improvement in Hypoglycemia Awareness
Description: Number of subjects with reduction of episodes of severe hypoglycemia and the presence of awareness of hypoglycemia
Time Frame: for the duration of islet graft function
Measure: Count of Participants; unit: Participants
Arm/Group | Islet Transplantation and Bone Marrow
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Arm/Group | Islet Transplantation and CD34 Bone Marrow
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Islet Transplantation and CD34 Bone Marrow (N=3)
Syncope leading to fracture of Humerus (Cardiac disorders) | 1 (1)
Severe hypoglycemia (Endocrine disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Islet Transplantation and CD34 Bone Marrow (N=3)
Anxiety (Nervous system disorders) | 1 (1)
Tremors (Nervous system disorders) | 1 (2)
Insomina (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Retinal Hemorrhage (Eye disorders) | 1 (1)
Pruritic Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Facial Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Onychomycosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus in perianal area (Skin and subcutaneous tissue disorders) | 1 (1)
Neck rash non-pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (3)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Calf pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Left arm pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Oral ulcers (Gastrointestinal disorders) | 2 (3)
Nausea and vomiting (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Explosive Diarrhea (Gastrointestinal disorders) | 1 (1)
Gallbladder Thickening (Hepatobiliary disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (2)
Pretibial and ankle edema (Blood and lymphatic system disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (2)
Vasovagal reaction during procedure (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Severe Hypoglycemia (Endocrine disorders) | 1 (1)
High CPK (Metabolism and nutrition disorders) | 1 (2)
Elevated LFT (Metabolism and nutrition disorders) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
HPV infection (Infections and infestations) | 1 (1)
Cervical intraepithelial neoplasia (Reproductive system and breast disorders) | 1 (1)
Cervical Polyp (Reproductive system and breast disorders) | 1 (1)
Pharyngitis and Bronchitis (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (3)
Upper respiratory infection (Infections and infestations) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Candidiasis (Infections and infestations) | 1 (1)
Ringworm infection (Infections and infestations) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes